CLINICAL TRIAL: NCT02195414
Title: Clinical Evaluation of a Bioresorbable Sirolimus-eluting Coronary Scaffold in the Treatment of Patients With de Novo Coronary Artery Lesion (NeoVas): a First-in-Man Study
Brief Title: NeoVas Bioresorbable Coronary Scaffold First-in-Man Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lepu Medical Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPM-201401
Record Dates: First submitted 2014-07-16; First posted 2014-07-21 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-03

CONDITIONS: Coronary Artery Disease
Keywords: NeoVas; Bioresorbable scaffold; Sirolimus; First-in-Man
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NeoVas BCS (Experimental): The NeoVas sirolimus-eluting bioresorbable coronary scaffold system is a PLLA-based polymer scaffold and contains the antiproliferative drug sirolimus.
  Interventions: Device: NeoVas BCS

INTERVENTIONS:
Device: NeoVas BCS — The NeoVas First-in-Man study is a prospective, two centers, single arm trial, which will enroll a total of 30 patients. The hypothesis of this study is to evaluate clinical feasibility, safety, and efficacy of NeoVas sirolimus-eluting bioresorbable coronary scaffold in the treatment of patients with de novo coronary lesion. The primary endpoint is a composite endpoint of cardiac death, target vessel related myocardial infarction, and ischemia driven target lesion revascularization (TLF) at 1 month follow up. At 6 months, 1, 2, 3, 4 and 5 years follow-up, clinical endpoints include TLF (its individual components), Patient-oriented cardiac event (all cause death, all MI, and all revascularization) target vessel revascularization, scaffold thrombosis.
  Other Names: NeoVas bioresorbable coronary scaffold

SUMMARY:
The NeoVas First-in-Man study is a prospective, two centers, single arm trial, which will enroll a total of 30 patients. The hypothesis of this study is to evaluate clinical feasibility, safety, and efficacy of NeoVas sirolimus-eluting bioresorbable coronary scaffold in the treatment of patients with de novo coronary lesion.

DETAILED DESCRIPTION:
The primary endpoint is a composite endpoint of cardiac death, target vessel related myocardial infarction, and ischemia driven target lesion revascularization (TLF) at 1 month follow up. At 6 months, 1, 2, 3, 4 and 5 years follow-up, clinical endpoints include TLF (its individual components), Patient-oriented cardiac event (all cause death, all MI, and all revascularization) target vessel revascularization, scaffold thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Age must be between 18 and 75 years, men or unpregnant women
* Patient must have evidence of myocardial ischemia (e.g., stable angina, unstable angina)
* Total number of target lesion =1 per patient
* Target lesion must be ≤ 20mm in length (visual estimation) and 2.75 to 3.75 mm in diameter（Online QCA）
* Target lesion is with a visually estimated stenosis of ≥ 70% (or ≥50% and evidence of myocardial ischemia) with a TIMI flow of ≥ 1
* The target lesion can be covered by one scaffold
* Patient must be an acceptable candidate for coronary artery bypass graft.
* Patient is able to verbally confirm understanding of risks, benefits and treatment of receiving the NeoVas bioresorbable coronary scaffold and he/she or his/her legally authorized representative provides written informed consent prior to any clinical investigation related procedure, as approved by the appropriate Ethics Committee of the respective clinical site.

Exclusion Criteria:

* Patients has had a known diagnosis of acute myocardial infarction (AMI) within 30 days preceding the procedure; CK and CK-MB have not returned within normal limits at the time of procedure
* Chronic total occlusion lesions(TIMI 0 grade blood flow prior to implantation), left trunk vessel lesion, ostial lesion ,multi-branch lesions needing treated, fork and bridge vessel lesions of branch vessels whose diameter ≥2.0mm(branch opening stenosis exceeds 40% or need balloon expansion); there is thrombus visible in the target blood vessels.
* Severe calcified lesions and twisted lesions which cannot be pre-expanded, and lesions unsuitable for delivering and expanding stents
* In-stent restenosis lesion
* Patient has undergone previous stenting anywhere within the target vessel(s) within the previous 12 months, or will require stenting within the target vessel(s) within 6 months after the study procedure; target vessels that has been planted stents over a year.
* Severe heart failure(over NYHA III grade ), or left ventricular ejection fraction(LVEF)< 40%( supersonic inspection or left ventricular radiography )
* Known renal insufficiency (e.g., eGFR <60 ml/min, or subject on dialysis)
* Patients with hemorrhage tendency, an active digestive ulcer history, a cerebral hemorrhage or subarachnoid hemorrhage history, or cerebral apoplexy within half a year, and these patients who contraindicate against platelet inhibitors and anticoagulant therefore can not bear anticoagulation treatment
* Patient has a known hypersensitivity or contraindication to aspirin, clopidogrel, heparin, contrast agent, polylactic acid or sirolimus that cannot be adequately pre-medicated
* Life expectancy < 12 months
* Patient is participating in another device or drug study that has not reached the primary endpoint of the study.
* Patient's inability to fully cooperate with the study protocol which in the investigator's opinion may limit his/her ability to participate in the study
* Patient has a heart transplant.
* Patient has current unstable arrhythmias, such as high risk ventricular premature beat and ventricular tachycardia.
* Patient is receiving or scheduled to receive chemotherapy for malignancy within 30 days prior to or after the procedure
* Patient is receiving immunosuppression therapy and has known immunosuppressive or autoimmune disease
* Patient is receiving or scheduled to receive chronic anticoagulation therapy (e.g., heparin, coumadin)
* Elective surgery is planned within the first 6 months after the procedure that will require discontinuing either aspirin or clopidogrel
* Platelet count <100,000 cells/mm3 or >700,000 cells/mm3, a WBC of <3,000 cells/mm3, or documented or suspected liver disease (including laboratory evidence of hepatitis)
* Patient has extensive peripheral vascular disease that precludes safe 6 French sheath insertion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-07; Primary Completion 2014-11 (Actual); Study Completion 2019-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, MD, Study Chair — The general hospital of Shenyang military region; Guosheng Fu, Principal Investigator — Sir Run Run Shaw Hospital; Bo Xu, Principal Investigator — Beijing Fuwai hospital, National center for cardiovascular diseases China; Yao-Jun Zhang, PhD, Principal Investigator — Nanjing First Hospital, Nanjing Medical University
Locations (2):
- China (2):
  - The General Hospital of Shenyang Military Region, Shenyang, Liaoning
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled into this trial were comprised of male and female subjects from the general interventional cardiology population. The study commenced on June 19, 2014 with the first subject enrolled on this date. The last subject was enrolled September 3, 2014.
Groups:
- NeoVas BCS: Patients received the NeoVas sirolimus-eluting bioresorbable coronary scaffold system, which is a PLLA-based polymer scaffold and contains the antiproliferative drug sirolimus.
Period: Overall Study
Arm/Group | NeoVas BCS
Started | 31
Primary Endpoint | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | NeoVas BCS
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] — Age must be between 18 and 75 years.
  years | 59.1 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 24
Diabetes Mellitus [Number; unit: participants]
  Yes | 7
  No | 24
Hypertension [Number; unit: participants]
  Yes | 16
  No | 15
Angina Categories [Number; unit: participants]
  Stable angina | 7
  Unstable angina | 23
  NSTEMI | 1
Target vessel location [Number; unit: participants]
  Left anterior descending artery | 17
  Left circumflex artery | 3
  Right coronary artery | 11
Stent diameter [Mean (Standard Deviation); unit: millimeter] | 3.35 (0.23)
Stent length [Mean (Standard Deviation); unit: millimeter] | 19.35 (3.54)

OUTCOME MEASURES:

1. Primary Outcome: Target Lesion Failure(TLF)
Description: Target lesion failure is a composite endpoint of cardiac death, target vessel related myocardial infarction (TV-MI) and the ischemia-driven target lesion revascularization.
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | NeoVas BCS
Number analyzed (Participants) | 31
participants
  Yes | 0
  No | 31

2. Secondary Outcome: Target Lesion Failure
Description: as for outcome 1
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2016-04

3. Secondary Outcome: Target Lesion Failure
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2016-10

4. Secondary Outcome: Target Lesion Failure
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2017-10

5. Secondary Outcome: Target Lesion Failure
Time Frame: 3 years
Reporting Status: Not Posted, anticipated posting 2018-10

6. Secondary Outcome: Target Lesion Failure
Time Frame: 4 years
Reporting Status: Not Posted, anticipated posting 2019-10

7. Secondary Outcome: Target Lesion Failure
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2020-10

8. Secondary Outcome: Patient Oriented Composite Endpoint
Description: Patients oriented composite endpoint includes all-cause death, all myocardial infarction and any revascularization.
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | NeoVas BCS
Number analyzed (Participants) | 31
participants | 0

9. Secondary Outcome: Patient Oriented Composite Endpoint
Description: Patients oriented composite endpoint includes all-cause death, all myocardial infarction and any revascularization.
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2016-04

10. Secondary Outcome: Patient Oriented Composite Endpoint
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2016-10

11. Secondary Outcome: Patient Oriented Composite Endpoint
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2016-10

12. Secondary Outcome: Patient Oriented Composite Endpoint
Time Frame: 3 years
Reporting Status: Not Posted, anticipated posting 2017-10

13. Secondary Outcome: Patient Oriented Composite Endpoint
Time Frame: 4 years
Reporting Status: Not Posted, anticipated posting 2018-10

14. Secondary Outcome: Patient Oriented Composite Endpoint
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2019-10

15. Secondary Outcome: Acute Success (Clinical Device and Clinical Procedure)
Description: Successful delivery and deployment of the Clinical Investigation scaffold at the intended target lesion and successful withdrawal of the scaffold delivery system with attainment of final residual stenosis of less than 50% of the target lesion by QCA (by visual estimation if QCA unavailable).
  Successful delivery and deployment of the Clinical Investigation scaffold at the intended target lesion and successful withdrawal of the scaffold delivery system with attainment of final residual stenosis of less than 50% of the target lesion by QCA (by visual estimation if QCA unavailable) and/or using any adjunctive device without the occurrence of ischemia driven major adverse cardiac event (MACE) during the hospital stay with a maximum of first seven days post index procedure. In dual lesion setting both lesions must meet clinical procedure success.
Time Frame: acute
Measure: Number; unit: participants
Arm/Group | NeoVas BCS
Number analyzed (Participants) | 31
participants
  Success | 31
  Failure | 0

16. Secondary Outcome: Scaffold Thrombosis
Description: Scaffold thrombosis will be categorized as acute (≤1day), subacute (>1day ≤30 days) and late (>30 days).
  Clinical presentation of acute coronary syndrome with angiographic evidence of scaffold thrombosis (angiographic appearance of thrombus within or adjacent to a previously treated target lesion).
  In the absence of angiography, any unexplained death, or acute MI (ST segment elevation or new Q-wave)* in the distribution of the targetlesion within 30 days.
Time Frame: 30days
Measure: Number; unit: participants
Arm/Group | NeoVas BCS
Number analyzed (Participants) | 31
participants | 0

17. Secondary Outcome: Scaffold Thrombosis
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2016-04

18. Secondary Outcome: Scaffold Thrombosis
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2016-10

19. Secondary Outcome: Scaffold Thrombosis
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2017-10

20. Secondary Outcome: Scaffold Thrombosis
Time Frame: 3 years
Reporting Status: Not Posted, anticipated posting 2018-10

21. Secondary Outcome: Scaffold Thrombosis
Time Frame: 4 years
Reporting Status: Not Posted, anticipated posting 2019-10

22. Secondary Outcome: Scaffold Thrombosis
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2020-10

23. Secondary Outcome: Angiographic Endpoint
Description: In-segment In-scaffold, proximal and distal Late lumen loss (mm); In-segment In-scaffold, proximal and distal Minimal lumen diameter(mm); In-segment In-scaffold, proximal and distal Diameter stenosis (%) Angiographic Binary Restenosis (%).
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2016-04

24. Secondary Outcome: Angiographic Endpoint
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2016-10

25. Secondary Outcome: Angiographic Endpoint
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2020-10

26. Secondary Outcome: OCT Endpoint
Description: proportion of covered struts, malapposed struts; neointimal hyperplasia (NIH) area, volume; NIH volume obstruction.
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2016-04

27. Secondary Outcome: OCT Endpoint
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2017-10

28. Secondary Outcome: OCT Endpoint
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2020-10

29. Secondary Outcome: IVUS Endpoint
Description: mean/minimal vessel area, mean/minimal lumen area, mean/minimal stent area
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2016-04

30. Secondary Outcome: IVUS Endpoint
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2017-10

31. Secondary Outcome: IVUS Endpoint
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2020-10

32. Secondary Outcome: MSCT Endpoint
Description: mean/minimal vessel area, mean/minimal lumen area, mean/minimal stent area
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2016-10

33. Secondary Outcome: MSCT Endpoint
Time Frame: 3 years
Reporting Status: Not Posted, anticipated posting 2018-10

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | NeoVas BCS
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No